CLINICAL TRIAL: NCT06295315
Title: Evaluation of the Psychological Profile of Adult Patients With Prader-Willi Syndrome
Acronym: PROPSICOPWS
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 01C310
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willy syndrome; Psychological well-being; Quality of life; Psychological distress
MeSH Terms: conditions — Prader-Willi Syndrome; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The primary aim of the present study is to investigate the psychological profile of adult patients with PWS and the fatigue experienced by family members. Specifically, the level of psychological well-being, the subjective perception of life quality, and the main characteristics present in terms of psychopathological functioning of subjects with PWS will be investigated. These variables will be investigated in order to detect their presence and the main bonds of interaction, either between them or with other socio-demographic data, in a sample of adults with PWS. At the same time, the presence of psychological distress, levels of well-being quality of life, and coping strategies in family members and caregivers of individuals with PWS will be investigated.

DETAILED DESCRIPTION:
The observational study will be carried out at the U.O. of Auxology, Istituto Auxologico Italiano, IRCCS, Piancavallo.

36 subjects with a genetic diagnosis of PWS, of both sexes and aged between 18 and 55, and their caregivers will be taken into consideration.

In subjects affected by PWS, the following variables will be investigated:

* anthropometric parameters (height, weight, BMI, waist circumference);
* socio-demographic conditions (gender, age, origin, level of education, family composition)
* concomitant hormonal and psychiatric therapies
* intellectual profile through the Mini-Mental State Examination (MMSE), a neuropsychological test consisting of 30 items that refer to the following cognitive areas: orientation in time, orientation in space, word recording, attention and calculation, recall, language, constructional praxis.
* psychological well-being through the Psychological General Well-Being Index (PGWBI), a questionnaire made up of 22 items that measure the following dimensions: anxiety, depression, positivity and well-being, self-control, general state of health, and vitality.
* perception of life quality through the 36-Item Short Form Survey (SF-36), a questionnaire composed of 36 items that investigates the perception of quality of life in relation to: physical functioning, limitations due to physical health, limitations due to emotions, energy and fatigue, emotional well-being, social activities, pain, general health perception
* mental distress through the Symptom Checklist-90-R (SCL-90-R), a questionnaire made up of 90 items capable of investigating the presence and severity of symptoms of mental distress related to nine psychopathological dimensions: somatization, obsession-compulsion, interpersonal sensitivity, depression, anxiety, anger-hostility, phobic anxiety, paranoid ideation, psychoticism.

The following variables will be investigated in the parents or caregivers of subjects with PWS:

* psychological distress through the Depression, Anxiety, and Stress Scale (DASS-21), a questionnaire composed of 21 items aimed at investigating experiences of anxiety, depression, and stress
* psychological well-being through the Psychological General Well-Being Index (PGWBI), a questionnaire made up of 22 items that measure the following dimensions: anxiety, depression, positivity and well-being, self-control, general state of health, and vitality.
* coping strategies through Coping Orientation to Problem Experienced (COPE-new Italian version). It is a questionnaire made up of 60 items aimed at investigating how often the subject implements - in difficult or stressful situations - different coping strategies to deal with stressful daily situations.
* hyperphagia of subjects with PWS through the Hyperphagia Questionnaire (HQ), a questionnaire to be administered to parents or caregivers of reference consisting of 11 items capable of investigating the hyperphagia of subjects affected by PWS.

ELIGIBILITY:
Inclusion Criteria: subjects with a genetic diagnosis of PWS capable of understanding the questionnaires

Exclusion Criteria: subjects with a genetic diagnosis of PWS with cognitive problems (evaluated throughout the Mini-Mental State Examination)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects with a genetic diagnosis of PWS, hospitalized at the Division of Auxology, Istituto Auxologico Italiano, Piancavallo-Verbania (Italy) for a 3-week body weight reduction program
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Psychological well-being through the Psychological General Well-Being Index (PGWBI) | Baseline
  A neuropsychological test consisting of 30 items that refer to the following cognitive areas: orientation in time, orientation in space, word recording, attention and calculation, recall, language, constructional praxis.
Perception of life quality through the 36-Item Short Form Survey (SF-36) | Baseline
  A questionnaire composed of 36 items that investigates the perception of quality of life in relation to: physical functioning, limitations due to physical health, limitations due to emotions, energy and fatigue, emotional well-being, social activities, pain, general health perception
Mental distress through the Symptom Checklist-90-R (SCL-90-R) | Baseline
  A questionnaire made up of 90 items capable of investigating the presence and severity of symptoms of mental distress related to nine psychopathological dimensions: somatization, obsession-compulsion, interpersonal sensitivity, depression, anxiety, anger-hostility, phobic anxiety, paranoid ideation, psychoticism.

SECONDARY OUTCOMES:
Psychological distress through the Depression, Anxiety, and Stress Scale (DASS-21) | Baseline (investigated in the parents or caregivers of subjects with PWS)
  A questionnaire composed of 21 items aimed at investigating experiences of anxiety, depression, and stress
Coping strategies through Coping Orientation to Problem Experienced (COPE-new Italian version). | Baseline (investigated in the parents or caregivers of subjects with PWS)
  A questionnaire made up of 60 items aimed at investigating how often the subject implements - in difficult or stressful situations - different coping strategies to deal with stressful daily situations.
Hyperphagia of subjects with PWS through the Hyperphagia Questionnaire (HQ) | Baseline (investigated in the parents or caregivers of subjects with PWS)
  A questionnaire to be administered to parents or caregivers of reference consisting of 11 items capable of investigating the hyperphagia of subjects affected by PWS.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, site Piancavallo, Oggebbio, Verbania, Italy